CLINICAL TRIAL: NCT05845827
Title: Impact of Dietary Intake on Continuous Glucose Patterns Considering Cardiorespiratory Fitness Levels.
Brief Title: Dietary Impact on Continuous Glucose Monitoring
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Jennifer L. Meijer, Assistant Professor of Medicine, Dartmouth-Hitchcock Medical Center
Other Study IDs: STUDY02001962
Record Dates: First submitted 2023-04-14; First posted 2023-05-06 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Glucose Metabolism Disorders; Dietary Habits; Pediatric ALL; Adult ALL
MeSH Terms: conditions — Glucose Metabolism Disorders; Feeding Behavior; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and buffy coat will be extracted from one blood sample (10mL).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiorespiratory fitness (CRF), also known as "exercise capacity", is the capacity of respiratory and circulatory systems to supply oxygen to skeletal muscle during exercise for the generation of energy. Determinants of CRF include lung capacity, capillary density, cardiac output, hemoglobin concentration, and mitochondrial function. The research group studies how CRF is related to fuel utilization, yielding a mechanistic understanding of the association between lower CRF and worsening metabolic health via mitochondrial function. The objective of this study is to measure fuel utilization in response to habitual diet for one week in adolescents and young adults, ages 14-22 years (n=30). Fuel utilization will be estimated by glucose measures using a continuous glucose monitor (CGM). Habitual dietary intake will be collected via a mobile phone application (BiteAI, Inc) that uses artificial intelligence to extract nutrient information from food photographs. Participants will undergo two standard of care (SOC) meal tolerance tests at home - a glucose tolerance test and a Ensure® mixed meal tolerance test. CRF will be estimated by measuring maximum oxygen consumption (VO2 max) during a graded treadmill test. The hypothesis is that a higher VO2 max will be associated with increased fuel utilization, measured by lower glucose response to the SOC meal tolerance tests. The proposed study is described in the following aims:

SPECIFIC AIM 1. Test for feasibility of completion of self-report dietary food records, completion of two at home meal tolerance tests that are standard of care for metabolic health screening, and completion of a seven-day continuous glucose monitor.

SPECIFIC AIM 2. Identify nutrients and foods that are associated with an elevated glucose response.

SPECIFIC AIM 3. Assess the influence of VO2 max on the glucose response to the SOC glucose tolerance test and Ensure® mixed meal tolerance test.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and young adults, ages 14-22 years

Exclusion Criteria:

* Previous diagnosis of type 1 or 2 diabetes
* Previous diagnosis of hyperlipidemia or other metabolic disease
* Use of medications known to affect glucose metabolism (metformin, oral steroids, sulfonylureas, insulin).
* Allergies to milk.
* Inability to participant in the maximal exercise test on the treadmill.
* Individuals not having android or IOS phones
* Individuals who cannot speak and/or write in English.

Ages: 14 Years to 22 Years | Sex: All
Age Groups: Child, Adult
Study Population: Adolescents and young adults, ages 14-22 years
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Number of dietary records completed by each study participant | 7-10 days
  The researchers will measure dietary intake using a mobile phone application called BiteSnap. The goal is to have participants report >90% of their meals using mobile phone photos to extract nutrient information.
Number of days wearing the continuous glucose monitor | 7-10 days
  The researchers will measure the amount of time each participant wears the continuous glucose monitor. The goal is to have participants wear the monitor for >90% of the time in the study.
Completion of the at-home glucose tolerance test | 7-10 days
  Participants will be asked to drink a 75-gram glucose tolerance test. The researchers will measure the number of participants that self-reported drinking the shake at fasting. The goal will be 90% of participants self-report drinking the shake at fasting.

SECONDARY OUTCOMES:
Identify nutrients associated with an elevated glucose response, measured by the continuous glucose monitor. | 7-10 days
  Participants will track the foods they eat while wearing the Dexcom continuous glucose monitors. Researchers will identify specific foods that are associated with increases in glucose response, considering associations across the group and associations within each individual.
Access the relationship between fitness levels and glucose response to standard of care meal tests. | 7-10 days
  Researchers will assess the association between fitness levels and glucose levels at 60 and 120 minutes after the at-home standard of care meal tests. Fitness levels are measured using a VO2 max test.

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ge M, Lebby SR, Chowkwale S, Harrison C, Palmer GM, Loud KJ, Gilbert-Diamond D, Vajravelu ME, Meijer JL. Impact of Dietary Intake and Cardiorespiratory Fitness on Glycemic Variability in Adolescents: An Observational Study. Curr Dev Nutr. 2025 Jan 21;9(2):104547. doi: 10.1016/j.cdnut.2025.104547. eCollection 2025 Feb. PMID 39996052